CLINICAL TRIAL: NCT04735796
Title: A Phase I, First-in-Human, Open-Label, Dose Escalation Study of LM-102 Injection in Subjects With CLDN18.2-Positive Advanced Solid Tumors
Brief Title: Study of LM-102 in Subjects in Advanced Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business strategy changed
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: LM102-01-101
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Dose level 1: 3mg/kg, enroll CLDN18.2 positive advanced solid tumors
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LM102 Dose Escalation Level 1, 3mg/kg (Experimental): LM102 Dose Escalation Level 1, 3mg/kg, enrolled CLDN 18.2 positive advanced solid tumors
  Interventions: Drug: Drug：LM-102
- LM102 Dose Escalation Level 2, 10mg/kg (Experimental): LM102 Dose Escalation Level 2, 10mg/kg,enrolled CLDN 18.2 positive advanced solid tumors
  Interventions: Drug: Drug：LM-102
- LM102 Dose Escalation Level 3, 20mg/kg (Experimental): LM102 Dose Escalation Level 3, 20mg/kg,enrolled CLDN 18.2 positive advanced solid tumors
  Interventions: Drug: Drug：LM-102
- LM102 Dose Escalation Level 4, 30mg/kg (Experimental): LM102 Dose Escalation Level 4, 30mg/kg,enrolled CLDN 18.2 positive advanced solid tumors
  Interventions: Drug: Drug：LM-102
- LM102 Dose Escalation Level 5, 40mg/kg (Experimental): LM102 Dose Escalation Level 5, 40mg/kg,enrolled CLDN 18.2 positive advanced solid tumors
  Interventions: Drug: Drug：LM-102

INTERVENTIONS:
Drug: Drug：LM-102 — Traditional '3+3' escalation design will be used. Dose escalation consists of five ascending dose levels of LM-102 (3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg and 40 mg/kg). All subjects will be administered every 3 weeks (1 cycle=21 days) with a dose of LM-102 as a 2 h (120±10 min) intravenous (IV) infusion until the disease progression, intolerance, subject discontinuation/informed consent withdrawal, or at the discretion of the investigator in consultation with sponsor, at most till by one year.

SUMMARY:
This is a phase Ⅰ, first-in-human, open-label, dose escalation study to evaluate the safety and tolerability, PK, immunogenicity and preliminary anti-tumor activity of LM-102 injection in subjects with CLDN18.2-positive advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase Ⅰ, first-in-human, open-label, dose escalation study to evaluate the safety and tolerability, PK, immunogenicity and preliminary anti-tumor activity of LM-102 injection in subjects with CLDN18.2-positive advanced solid tumors.

Dose Escalation Traditional '3+3' escalation design will be used. Dose escalation consists of five ascending dose levels of LM-102 (3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg and 40 mg/kg). All subjects will be administered every 3 weeks (1 cycle=21 days) with a dose of LM-102 as a 2 h (120±10 min) intravenous (IV) infusion until the disease progression, intolerance, subject discontinuation/informed consent withdrawal, or at the discretion of the investigator in consultation with sponsor.

After all the subjects in each cohort complete the DLT assessment, the safety monitor committee (SMC) will make decisions for dose escalations, exploring intermediate/higher doses or terminating dose escalations according to the safety, tolerability, PK and immunogenicity data. The SMC may also adjust the dosage, frequency of administration, PK sample collection plan, etc.

Based upon safety, tolerability, PK, and immunogenicity, the MTD or OBD will be determined by SMC. And the RP2D will be determined based on DLTs, MTD or OBD, and the totality of the safety data throughout the study, including dose modifications and delays, PK, and immunogenicity data, etc.

The study will consist of 3 periods:

1. Screening period (up to 28 days before the first dose);
2. Treatment period;
3. Follow-up period [28 (±3) days after end of treatment (EOT)/early withdrawal or before other anti-tumor treatments (whichever occurs earlier)].

Safety, tolerability and anti-tumor activity evaluation of LM-102 will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent document prior to any procedure; 2. Aged between 18 to 75 years old, male or female when sign the informed consent form (ICF); 3. Subjects must have histological or cytological confirmation of recurrent or refractory CLDN18.2-positive advanced solid tumors including but not limit to gastric and gastroesophageal junction adenocarcinoma, pancreatic carcinoma, biliary tract carcinoma, colorectal carcinoma, ovarian carcinoma; 4. Subjects are intolerable for available standard therapy or there is no standard available therapy; 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 with no deterioration within 2 weeks from the first dose; 6. Life expectancy ≥ 3 months; 7. Tumor samples have CLDN18.2 membranous staining in ≥ 1% of the tumor cells with any intensity as determined by central immunohistochemistry (IHC) testing. As such, all patients must be able to provide formalin fixed and paraffin embedded archived tumor tissue samples obtained ≤ 3 years prior to screening; 8. Subjects must have the following organ and marrow function in laboratory tests within 7 days from the first dose:

  1. PLT ≥ 90 × 109/L; ANC ≥ 1.5 × 109/L; Hemoglobin ≥ 9 g/dL, without receiving EPO, G-CSF, or GM-CSF within 14 days and blood transfusion in at least 7 days;
  2. Coagulation function: INR ≤ 1.5; APTT ≤ 1.5 × ULN;
  3. Liver function: Bilirubin ≤ 1.5 × ULN (Subjects with Gilbert's Syndrome are allowed if direct bilirubin is within normal limits); AST and ALT≤ 2.5 × ULN without liver metastases (≤ 5 × ULN if liver metastases are present); Albumin ≥ 2.5 g/dL;
  4. Kidney function: Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula, see Appendix 2); Qualitative urine protein ≤ 1+ or qualitative urine protein ≥ 2+, but 24-hour urine protein < 1g;
  5. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%, QT interval (QTcF) ≤ 470 ms.

     9. Subjects who are able to well communicate with investigators as well as understand and adhere to the requirements of this study.

     Exclusion Criteria:
     1. Subjects who have difficulties in venous blood collection or history of dizziness with blood or needles;
     2. Childbearing potential female (see Appendix 3 Contraceptive Methods) who have positive pregnancy test or are breast feeding;
     3. Subjects who known to be allergic to LM-102 or any of its excipients;
     4. Exposure to any IMP, or participate in any other clinical trial within 28 days prior to 1st dosing LM-102;
     5. Subjects with prior anti-tumor within 28 days prior to 1st dosing of LM-102, including radiotherapy (except palliative radiotherapy, beyond 14 days prior to 1st dosing of LM-102, and the toxicity has been recovered as assessed by investigator.), chemotherapy, biotherapy, endocrine therapy and immunotherapy, etc. However, the application of other small molecular targeted drugs and the herbal medicine with anti-tumor indication longer than 14 days or 5 half-life periods of the drug (whichever is longer) is acceptable;
     6. Subjects who have received surgical or interventional treatment within 28 days prior to 1st dosing LM-102, excluding operations or surgeries that can be recovered within 14 days prior to 1st dosing LM-102, and have been recovered by the investigator's assessment, e.g., tumor biopsy, puncture, palliative operation, rectal/gastrostomy, etc.;
     7. Subjects who have concurrent administration of anticoagulation agents or vitamin K antagonists;
     8. Subjects who have concurrent administration of therapeutic doses of heparin (prophylactic doses are acceptable);
     9. Subjects who have gastric outlet obstruction, persistent recurrent vomiting or uncontrolled/significant gastrointestinal hemorrhage, symptomatic peptic ulcer, or major bleeding risk in other parts of the body within 28 days prior to 1st dosing LM-102;
     10. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence that the subject's central nervous system metastasis or meningeal metastasis has not been controlled, and the investigator judges it to be unsuitable for inclusion;
     11. Subjects who have symptomatic congestive heart failure, history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina pectoris, uncontrolled hypertension (Blood pressure still ≥ 140/90 mmHg after drug treatment), clinically significant cardiac arrhythmia or myocardial infarction within the past 6 months, etc.;
     12. Any adverse events from prior anti-tumor therapy have not yet recovered to ≤ grade 1 of CTCAE v5.0 (Except for some grade 2 toxicity that the investigator judges that there is no safety risk, such as alopecia, and other long term ≤ grade 2 toxicities which would not impact the administration of LM-102 and safety evaluation);
     13. Subjects who have uncontrolled or severe illness, including but not limited to ongoing or active infection requiring antibiotics;
     14. Subjects who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation, or allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
     15. HIV infection, active HBV infection (HBV DNA exceeds the ULN), active HCV infection (HCV RNA exceeds the ULN);
     16. Male and female subjects who are unwilling to use adequate contraceptive methods (e.g, concomitant use of a spermicidal agent, barrier contraceptive, or/and intrauterine contraceptive during the study and for at least 6 months after the last dose of LM-102. (See Appendix 3 for contraceptive methods);
     17. Subjects who have psychiatric illness or social situations that would preclude study compliance;
     18. Subjects who have another active malignancy which is likely to require treatment;
     19. Subject who is determined as not eligible to participate in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | From screening up to 1 year
  The safety profile of LM102 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Maximum tolerated dose (MTD) | Cycle 1 of each cohort. Duration of one cycle is 3 weeks
  MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycle
Dose-limiting toxicities (DLT) | Cycle 1 of each cohort. Duration of one cycle is 3 weeks
  DLT is defined as a toxicity (adverse event at least possibly related to YH002) occurring during the DLT observation period (the initial 21 days)
Change in Vital Signs-ear temperature | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Change in vital signs-ear temperature will be measured after the subject has been fully rested.
Change in Vital Signs-pluse rate | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Change in vital signs-pluse rate will be measured after the subject has been fully rested.
Change in Vital Signs-blood pressure | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Change in vital signs-blood pressure will be measured after the subject has been fully rested.
Change in Electrocardiogram (ECG)-RR interval | Baseline (Week 0) through approximately 1 year after first administration of LM102
  RR interval of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once. RR is the standard heart rate which calculated by 60 divided by heart rate.
Change in Electrocardiogram (ECG)-QT interval | Baseline (Week 0) through approximately 1 year after first administration of LM102
  QT interval of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once.
Change in Electrocardiogram (ECG)-QRS duration | Baseline (Week 0) through approximately 1 year after first administration of LM102
  QRS duration of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once.
Incidence of Abnormal Clinical Laboratory Test Results-hematology | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Number of participants with incidence of abnormal clinical lab test results like hematology will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Biochemistry | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Number of participants with incidence of abnormal clinical lab test results like Biochemistry will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Urinalysis | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Number of participants with incidence of abnormal clinical lab test results like Urinalysis will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Coagulation test | Baseline (Week 0) through approximately 1 year after first administration of LM102
  Number of participants with incidence of abnormal clinical lab test results like Coagulation test will be assessed.

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve within one dosing interval (AUCtau) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM102
Volume of distribution (Vd) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM102
Volume of distribution at steady state (Vss) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM102
Maximum serum concentration (Cmax) | Up to 1 year
  To determine the PK profile of LM102 as single agent
Trough concentration before the next dose is administered (Ctrough) | Up to 1 year
  To determine the PK profile of LM102
Time to reach maximum serum concentration (Tmax) | Up to 1 year
  To determine the PK profile of LM102
Clearance (CL) | Up to 1 year
  To determine the PK profile of LM102
Terminal half-life (T1/2) | Up to 1 year
  To determine the PK profile of LM102
Dose proportionality | Up to 1 year
  To determine the PK profile of LM102
Incidence of anti-drug antibodies (ADAs) | Up to 1 year
  To assess the immunogenicity of LM102
Incidence of neutralizing antibodies (NAbs) | Up to 1 year
  To assess the immunogenicity of LM102
Objective response rate (ORR) | Up to 1 year
  To assess the preliminary antitumor activity of LM102,The ORR, using RECIST 1.1 criteria, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) at any time during the study, based on Investigator assessment.
Best of response (BOR) | Up to 1 year
  To assess the preliminary antitumor activity of LM102
Disease control rate (DCR) | Up to 1 year
  To assess the preliminary antitumor activity of LM102

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sarcoma Oncology Research Center, Cancer Center of Southern California, California City, California
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Oklahoma University- Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Texas MD Anderson Cancer Center, Houston, Texas